CLINICAL TRIAL: NCT03646604
Title: An Open-label Multiple Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Upadacitinib in Pediatric Subjects With Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Upadacitinib in Pediatric Participants With Severe Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M16-049; 2018-004409-17 (EudraCT Number)
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis
Keywords: Upadacitinib; ABT-494; Atopic Dermatitis; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1; Cohort 1 (Experimental): Participants, 6 to <12 years of age, will receive low dose of upadacitinib.
  Interventions: Drug: Upadacitinib (ABT-494)
- Part 1; Cohort 2 (Experimental): Participants, 6 to <12 years of age, will receive high dose of upadacitinib.
  Interventions: Drug: Upadacitinib (ABT-494)
- Part 1; Cohort 3 (Experimental): Participants, 2 to <6 years of age, will receive low dose of upadacitinib.
  Interventions: Drug: Upadacitinib (ABT-494)
- Part 1; Cohort 4 (Experimental): Participants, 2 to <6 years of age, will receive high dose of upadacitinib.
  Interventions: Drug: Upadacitinib (ABT-494)
- Part 2 (Experimental): Eligible participants who completed Part 1 will receive weight-dependant low dose of upadacitinib.
  Interventions: Drug: Upadacitinib (ABT-494)

INTERVENTIONS:
Drug: Upadacitinib (ABT-494) — Upadacitinib will be administered orally.
  Other Names: ABT-494; RINVOQ

SUMMARY:
The objective of this study is to evaluate the safety, pharmacokinetics and tolerability of multiple doses of upadacitinib in pediatric participants with severe atopic dermatitis and to evaluate palatability of upadacitinib oral solution in pediatric participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with total body weight of 10 kilograms(kg) or higher at Baseline. Beginning with protocol version 6.0, only subjects 3 years of age and older will be enrolled for the remainder of this study.
* Diagnosed with atopic dermatitis (AD) with onset of symptoms at least 6 months prior to baseline.
* Meets Hanifin and Rajka criteria for AD.
* Diagnosed with active severe AD defined by Eczema Area Severity Index (EASI), Validated Investigator's Global Assessment (IGA) and body surface area (BSA).
* Documented history (within 12 months prior to the Baseline Visit) of inadequate response or intolerance to topical corticosteroids (TCS) and topical calcineurin inhibitor (TCI) OR for whom use of TCS and TCIs is otherwise medically inadvisable.

Exclusion Criteria:

* Prior exposure to Janus Kinase (JAK) inhibitor.
* Requirement of prohibited medications during the study.
* Current use of known moderate or strong inhibitors or inducers of drug metabolizing enzymes within 30 days prior to the first dose of study drug and through the end of Part 1 of the study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to 7 days
  It is defined as the maximum observed plasma concentration (Cmax) for upadacitinib.
Time to Maximum Observed Plasma Concentration (Tmax) | Up to 7 days
  It is defined as the time to maximum plasma concentration (Tmax) of upadacitinib.
Area under the plasma concentration-time curve within a dosing interval (AUCtau) | Up to 7 days
  The area under the plasma concentration-time curve (AUCtau) is a method of measurement of the total exposure of a drug in plasma.
Oral Clearance | Up to 7 days
  Clearance is defined the volume of plasma cleared of the drug per unit time.
Number of Participants With Treatment Emergent Adverse Events (TEAE) | Up to 2 years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events (TEAEs) are defined as any event that began or worsened in severity after the first dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- United States (15):
  - Beach Pediatrics /ID# 207834, Huntington Beach, California
  - Children's Hospital Los Angeles /ID# 206042, Los Angeles, California
  - Pediatric Skin Research, LLC /ID# 213468, Coral Gables, Florida
  - Rybear, Inc /ID# 231801, Fort Lauderdale, Florida
  - IACT Health-Columbus /ID# 216370, Columbus, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 206224, Chicago, Illinois
  - Dawes Fretzin, LLC /ID# 214958, Indianapolis, Indiana
  - Duplicate_Washington University of St. Louis /ID# 206972, St Louis, Missouri
  - University of New Mexico School of Medicine /ID# 206757, Albuquerque, New Mexico
  - Cincinnati Children's Hospital /ID# 207071, Cincinnati, Ohio
  - Oregon Medical Research Center /ID# 206226, Portland, Oregon
  - Penn State University and Milton S. Hershey Medical Center /ID# 207096, Hershey, Pennsylvania
  - Paddington Testing Co., Inc. /ID# 207079, Philadelphia, Pennsylvania
  - Arlington Research Center, Inc /ID# 222901, Arlington, Texas
  - West Virginia University Hospitals /ID# 206792, Morgantown, West Virginia
- Norway (2):
  - Haukeland University Hospital /ID# 210162, Bergen, Hordaland
  - Rikshospitalet OUS HF /ID# 210163, Oslo
- Alma M. Cruz Santana, MD-Private practice /ID# 214890, Carolina, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qian Y, Raymundo EM, Hao S, Unnebrink K, Levy GF, Teixeira HD, Chu AD, Zinn ZA, Paller AS, Liu W, Mohamed MF. Pharmacokinetics, Safety, Tolerability, and Exploratory Efficacy of Upadacitinib in Children with Severe Atopic Dermatitis. Clin Ther. 2024 Oct;46(10):733-741. doi: 10.1016/j.clinthera.2024.07.003. Epub 2024 Aug 13. PMID 39142926
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M16-049#additional-resources-section